CLINICAL TRIAL: NCT00307970
Title: The Impact of an Anti-static Valved-holding Chamber on Bioavailability of Inhaled Fluticasone Propionate in Young Children With Asthma
Brief Title: Impact of Anti-static Chamber/Mask
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 582-2002
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2004-06

CONDITIONS: Asthma
Keywords: fluticasone; asthma therapy; spacer inhaler; HFA-134a
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: HFA FP MDI
Device: conventional chamber/mask; anti-static chamber/mask

SUMMARY:
To compare lung delivery of fluticasone propionate delivered by HFA-pMDI, using a conventional polycarbonate of anti-static chamber/mask in a randomized crossover design in 1-6 year old children.

Hypothesis: Anti-static chamber/mask would increase the amount of inhaled corticosteroid delivered to young children who passively inhale and cannot breath hold.

DETAILED DESCRIPTION:
Objective -- to determine whether an anti-static chamber increases the one-hour steady-state fluticasone plasma concentration, which is an indirect measure of airway delivery and direct measure of systemic exposure. Twelve children 1-6 yrs with well-controlled persistent asthma were treated with HFA-FP pMDI, 2 actuations of 110 µg twice daily. The drug was administered by conventional polycarbonate or anti-static valved-holding chambers with masks in an unblinded, randomized, crossover manner each for at least three days. A blood sample was collected one hour after the last dose when adherence documented by electronic monitor was 100%. FP plasma concentrations were measured by liquid chromatography mass spectrometry assay. Results evaluated using regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* children 1-6 years old; adequately controlled persistent asthma; currently receiving FP delivered by CFC MDI attached to valved-holding chamber/mask; ability to use chamber with mask effectively

Exclusion Criteria:

* inadequately controlled asthma: nocturnal awakening > 2 nights/month, prn albuterol use > 2x/week, more than 2 short courses of oral corticosteroids in previous 3 months, missing a dose on more than one occasion, increase in asthma symptoms during study, inability to discontinue intranasal or dermal fluticasone for 3 days

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12
Dates: Start 2003-04; Study Completion 2003-09

PRIMARY OUTCOMES:
one-hour steady-state plasma concentration of fluticasone after each device

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Hendeles, PharmD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Asthma Research Lab, Gainesville, Florida, United States